CLINICAL TRIAL: NCT01847157
Title: The Effect of the Transcranial Direct Current Stimulation Combined Sensory Modulation Intervention on Upper Extremity Functional Rehabilitation in Patients With Chronic Stroke
Brief Title: Transcranial Direct Current Stimulation Combined Sensory Modulation Intervention in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201202016RIB
Record Dates: First submitted 2013-04-22; First posted 2013-05-06 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Stroke
Keywords: recovery of function; stroke; Upper extremity; Motor; transcranial direct current stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Lidocaine, Prilocaine Drug Combination; Lidocaine; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS & epidermis anesthesia & repeated passive movement (Experimental): The patients in the experiment group will receive multi-strategy combination treatment mode- "combined tDCS and sensory input regulation treatment mode", including bilateral tDCS , epidermis anesthesia in the proximal hand of affected side and in the distal hand of unaffected side , and repeated passive movement training for the hand of affected side.
  Treatment modes are 3 times a week, 30 minutes each time, lasting for 8 weeks, and totally 24 trainings. The treatment content of each strategy is separately described in the following.
  Interventions: Device: tDCS; Drug: Epidermis anesthesia; Other: Repeated passive movement
- Shame tDCS & sham anesthesia & repeated passive movement (Sham Comparator): the control group is "repeated passive movement stimulation", including sham bilateral tDCS, sham epidermis anesthesia in the proximal hand of affected side and in the distal hand of unaffected side, and repeated passive movement training for the hand of affected side.
  Treatment modes are 3 times a week, 30 minutes each time, lasting for 8 weeks, and totally 24 trainings. The treatment content of each strategy is separately described in the following.
  Interventions: Drug: sham anesthesia; Other: Repeated passive movement; Device: sham tDCS

INTERVENTIONS:
Device: tDCS — Intelect mobile combination (Intelect, USA) is utilized as a direct current stimulator. The 25 cm2 electrodes on a sponge slice immersed in physiological salt solution are fixed on the left and right positions C3/ C4 of subject head (according to the international 10-20 system of electroencephalogram).
  During the treatment, 1.5 mA electric current is applied to stimulate the subjects in the experimental group for totally 30 minutes. At the start and the end of stimulation, the electric current will gradually increase from zero, or reduce to zero in 1 minute in order to avoid the possible appearance of slight flash effect of subject eyesight, which is caused by instantly turning on or turning off the electric current.
  Other Names: Intelect mobile combination
  Arms: tDCS & epidermis anesthesia & repeated passive movement
Drug: Epidermis anesthesia — 15 g of Emla 5% Cream(anesthetic) is applied to the ventral surface of the forearm of unaffected side with a distance of 10 mm from the wrist, and an area of 150 mm long x 50 mm wide.
  Furthermore, 10 g Emla 5% Cream(anesthetic) is applied to the ventral surface of the upper arm of affected side with a distance of 10 mm from the wrist, and an area of 100 mm long x 50 mm wide.
  Other Names: Emla 5% cream (Lignocaine 2.5% / Prilocaine 2.5%)
  Arms: tDCS & epidermis anesthesia & repeated passive movement
Drug: sham anesthesia — 15 g of 5% body Cream is applied to the ventral surface of the forearm of unaffected side with a distance of 10 mm from the wrist, and an area of 150 mm long x 50 mm wide.
  10 g body Cream is applied to the ventral surface of the upper arm of affected side with a distance of 10 mm from the wrist, and an area of 100 mm long x 50 mm wide.
  Other Names: Cetaphil; body cream
  Arms: Shame tDCS & sham anesthesia & repeated passive movement
Other: Repeated passive movement — Repeated passive wrist extension training: Patients' wrist joint are passively moved by a trained occupational therapist (joint moving angle = 0- 60 degree), frequency 1 Hz, maintain for 20 minutes.
  Finger passive flexion and extension training: Patients' fingers joint are passively moved by a trained occupational therapist, frequency 1 Hz, maintain for 10 minutes.
Device: sham tDCS — The equipment of sham stimulation in the control group is exactly the same as the equipment in the experiment group. However, the only difference is that 30 seconds after the start of electric current, the experimenter turns off the powder under subject ignorance situation. The stimulation just gives patients weak sense of electric current, in order to blind them for which group they are in.
  Other Names: Intelect mobile combination
  Arms: Shame tDCS & sham anesthesia & repeated passive movement

SUMMARY:
Background and purpose:

About 30% of people with stroke suffered from severe long-term upper extremity （UE） motor impairment. Severe UE impairment, especially dysfunction of hand, can greatly impact stroke patients' daily living independence and quality of life. However, treatment effect of current interventions is still limited. Nick Ward and Leonardo Cohen suggested 5 intervention strategies for stroke motor recovery: （1） reduction of somatosensory input from the intact; （2） increase in somatosensory input from the paretic; （3） anesthesia of a body part proximal to the paretic hand; （4） activity within the affected motor cortex may be up-regulated; （5） activity within the intact motor cortex may be down-regulated. Recent studies have shown each strategy to be effective in stroke patients with mild or moderate UE impairment. However, evidence for people with severe UE impairment after stroke remains unclear. Since research has found a greater effect for combined strategies than a single strategy, this proposal develops a combined intervention with the above 5 strategies, named "transcranial direct current stimulation （tDCS） combined sensory modulation intervention". This intervention is expected to be most effective for people with severe UE impairment after stroke.

In addition, neuroimaging can provide in vivo information about the brain plasticity which underpinning the motor recovery after stroke. However, image indexes that can be used in stroke patients with severe UE impairment remained examined. Therefore, this proposal has 3 aims: （1） to examine the treatment effect of the "tDCS combined sensory modulation intervention" in stroke patients with severe UE impairment; （2） to examine the underline mechanism of the efficacy of "tDCS combined sensory modulation intervention" using neuroimaging technology.

Methods:

This study is a double-blinded randomized controlled trial which will recruit 60 people who have had stroke onset more than 6 months and have severe UE motor impairment. All participants will be randomly assigned into 2 groups. The experimental group will be given the "tDCS combined sensory modulation intervention", combining bilateral tDCS stimulation, anesthesia techniques and repetitive passive motor training. The control group is given sham tDCS, sham anesthesia and repetitive passive motor training. Each group will be evaluated for outcomes at 4 time points （i.e. baseline, post-intervention, 3 months and 6months post-intervention）. The immediate and long-term effect of the interventions will be examined.

Primary outcome indicators include upper extremity impairment measures. Secondary outcome measures include upper extremity function, activities of daily living function, functional Magnetic Resonance Imaging （fMRI）, and corticospinal tract structural integrity using diffusion spectrum imaging （DSI）. Fifteen subjects of each group will be assessed 2 times （i.e., prior to the intervention and after the intervention） for fMRI and DSI scan.

Anticipatory results and contributions:

The results of the studies are expected to present a potentially effective intervention for stroke patients with severe impaired UE motor. Imaging evidence of brain plasticity for this particular intervention is also provided. The results will contribute to our understanding of brain plasticity for UE motor recovery after stroke. Findings from this proposal may help researchers and clinicians choose or develop interventions that are optimal to their clients individually.

ELIGIBILITY:
Inclusion Criteria:

1. first ever ischemic or hemorrhagic stroke patients identified by computed tomography (CT) or magnetic resonance imaging (MRI)
2. age between 40 and 80 years old
3. have a stroke over 6 months
4. unilateral hemiplegia
5. Fugl-Meyer assessment-upper extremity (FMA-UE) score≦29 when selection
6. poststroke elbow flexor spasticity less than 2 using modified Ashworth scale (MAS)
7. no severe anesthesia (FMA sensory test, upper extremity score≧10 )
8. no wrist and finger joint pain
9. clear consciousness, can understand simple sentences and spoken orders, and co-operate manipulation
10. can accept motor training in the sitting position for approximately 30 minutes.

Exclusion Criteria:

1. Suffer from other orthopedic diseases (such as severe arthritis), nerve damage (such as peripheral nerve damage), or severe pain, which influences upper extremity motor
2. have a medical history or family history of epilepsy
3. regularly take central nervous system drugs (such as sedatives), or the Class III antiarrhythmic drugs (such as amiodarone)
4. have atopic dermatitis or skin disorders of the scalp
5. have allergy to anesthetic medicines of the acyl amine
6. have a metal implant in the head or neck, or serious arrhythmia (the heartbeat is less than 50 beats per minute or higher than 100 beats per minute); or use a pacemaker or atrial defibrillator
7. suffer from congenital or idiopathic methemoglobinemia. Aphasia is not an exclusion criterion, but the patients should understand simple spoken orders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline Fugl Meyer Assessment(FMA)upper extremities subscale after intervention | Assessed at the baseline section (within 3 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 3 days after the latest intervention section)
  FMA-UE estimates the movement of proximal upper extremity (including shoulder joint, elbow joint and forearm), wrist joint and hand.
  Each movement is estimated by 3 scaled rules (0-1-2): score 0 indicates that the patient has no movement at all; score 1 indicates that the patient can perform partial movements; score 2 indicates that the patient can normally perform all movements.
  The total score in the differential scale is 66, and a higher score indicates that the patient has better movement ability.
Change from baseline Active joint activity after intervention | Assessed at the baseline section (within 3 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 3 days after the latest intervention section)
  A protractor is used to estimate 4 active joint activities of patients,including wrist extension, carpometacarpal extension, metacarpophalangeal extension, and shoulder flexion.
Change from baseline Muscle tone after intervention | Assessed at the baseline section (within 3 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 3 days after the latest intervention section)
  Motor assessment scale (MAS) is used to estimate muscle tension in patients, and the estimated muscles include the flexors and extensors of elbow, wrist and metacarpophalangeal joints.
  MAS is totally divided into 6 scales (0, 1, 1+, 2, 3, 4), and a higher score indicates that the patient has higher muscle tension.

SECONDARY OUTCOMES:
Change from baseline research arm test (ARAT) after intervention | Assessed at the baseline section (within 3 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 3 days after the latest intervention section)
  ARAT measures 4 upper extremity functions, including grasp, grip, pinch, and gross motor. It includes 19 items using 4-point scale (0-1-2-3). Total score is 57.A higher score indicates that the patient has higher upper extremity function.
Change from baseline Barthel Index(BI) after intervention | Assessed at the baseline section (within 3 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 3 days after the latest intervention section)
  Barthel Index with total possible scores ranging from 0 to 20 is utilized to estimate patients' basic functions in daily life. It has 10 items. Higher scores indicate higher independence in daily life.
Change from baseline Patient Health Questionnaire (PHQ-9) after intervention | Assessed at the baseline section (within 3 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 3 days after the latest intervention section)
  PHQ-9 is used to evaluate patients' depressive symptoms. PHQ-9 includes 9 items, using 4-point scale (0-1-2-3) to estimate the appearance frequency of each depressive symptom. Total possible scores range from 0 to 27, and a higher score indicates a higher appearance frequency of melancholic symptoms.
Change from baseline fMRI activation after intervention | Assessed at the baseline section (within 3 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 3 days after the latest intervention section)
  3T Siemens whole body nuclear magnetic resonance imaging system (Trio, Siemens, Erlangen, Germany) with 32-channel phase-array head coil is utilized to collect image information.
  Patients put left and right hands in left and right pneumatic 10-finger stimulators (Mag Design and Engineering, USA), respectively. This instrument does not have any invasive risk.
Change from baseline Diffusion Spectrum Imaging after intervention | Assessed at the baseline section (within 7 days ahead to the 1st intervention section), and then again immediately following the 8 weeks intervention (within 7 days after the latest intervention section).
  3T Siemens whole body nuclear magnetic resonance imaging system (Trio, Siemens, Erlangen, Germany) with 32-channel phase-array head coil is utilized to collect image information.
  Patients are asked to lie down and keep relax on the scanning table for 20 minutes. This instrument does not have any invasive risk.
  Patients' corticospinal tract structural integrity will be analyzed after imaging preprocessing.
Change from baseline research arm test (ARAT) at 3 months after intervention | Assessed at 3 months after intervention
  ARAT measures 4 upper extremity functions, including grasp, grip, pinch, and gross motor. It includes 19 items using 4-point scale (0-1-2-3). Total score is 57.A higher score indicates that the patient has higher upper extremity function.
Change from baseline research arm test (ARAT) at 6 months after intervention | Assessed at 6 months after intervention
  ARAT measures 4 upper extremity functions, including grasp, grip, pinch, and gross motor. It includes 19 items using 4-point scale (0-1-2-3). Total score is 57.A higher score indicates that the patient has higher upper extremity function.
Change from baseline Barthel Index(BI) at 3 months after intervention | Assessed at 3 months after intervention
  Barthel Index with total possible scores ranging from 0 to 20 is utilized to estimate patients' basic functions in daily life. It has 10 items. Higher scores indicate higher independence in daily life.
Change from baseline Patient Health Questionnaire (PHQ-9) at 3 months after intervention | Assessed at 3 months after intervention
  PHQ-9 is used to evaluate patients' depressive symptoms. PHQ-9 includes 9 items, using 4-point scale (0-1-2-3) to estimate the appearance frequency of each depressive symptom. Total possible scores range from 0 to 27, and a higher score indicates a higher appearance frequency of melancholic symptoms.
Change from baseline Barthel Index(BI) at 6 months after intervention | Assessed at 6 months after intervention
  Barthel Index with total possible scores ranging from 0 to 20 is utilized to estimate patients' basic functions in daily life. It has 10 items. Higher scores indicate higher independence in daily life.
Change from baseline Patient Health Questionnaire (PHQ-9) at 6 months after intervention | Assessed at 6 months after intervention
  PHQ-9 is used to evaluate patients' depressive symptoms. PHQ-9 includes 9 items, using 4-point scale (0-1-2-3) to estimate the appearance frequency of each depressive symptom. Total possible scores range from 0 to 27, and a higher score indicates a higher appearance frequency of melancholic symptoms.
Change from baseline Fugl Meyer Assessment(FMA)upper extremities subscale at 3 months after intervention | Assessed at 3 months after intervention
  FMA-UE estimates the movement of proximal upper extremity (including shoulder joint, elbow joint and forearm), wrist joint and hand.
  Each movement is estimated by 3 scaled rules (0-1-2): score 0 indicates that the patient has no movement at all; score 1 indicates that the patient can perform partial movements; score 2 indicates that the patient can normally perform all movements.
  The total score in the differential scale is 66, and a higher score indicates that the patient has better movement ability.
Change from baseline Active joint activity at 3 months after intervention | Assessed at 3 months after intervention
  A protractor is used to estimate 4 active joint activities of patients,including wrist extension, carpometacarpal extension, metacarpophalangeal extension, and shoulder flexion.
Change from baseline Muscle tone at 3 months after intervention | Assessed at 3 months after intervention
  Motor assessment scale (MAS) is used to estimate muscle tension in patients, and the estimated muscles include the flexors and extensors of elbow, wrist and metacarpophalangeal joints.
  MAS is totally divided into 6 scales (0, 1, 1+, 2, 3, 4), and a higher score indicates that the patient has higher muscle tension.
Change from baseline Fugl Meyer Assessment(FMA)upper extremities subscale at 6 months after intervention | Assessed at 6 months after intervention
  FMA-UE estimates the movement of proximal upper extremity (including shoulder joint, elbow joint and forearm), wrist joint and hand.
  Each movement is estimated by 3 scaled rules (0-1-2): score 0 indicates that the patient has no movement at all; score 1 indicates that the patient can perform partial movements; score 2 indicates that the patient can normally perform all movements.
  The total score in the differential scale is 66, and a higher score indicates that the patient has better movement ability.
Change from baseline Active joint activity at 6 months after intervention | Assessed at 6 months after intervention
  A protractor is used to estimate 4 active joint activities of patients,including wrist extension, carpometacarpal extension, metacarpophalangeal extension, and shoulder flexion.
Change from baseline Muscle tone at 6 months after intervention | Assessed at 6 months after intervention
  Motor assessment scale (MAS) is used to estimate muscle tension in patients, and the estimated muscles include the flexors and extensors of elbow, wrist and metacarpophalangeal joints.
  MAS is totally divided into 6 scales (0, 1, 1+, 2, 3, 4), and a higher score indicates that the patient has higher muscle tension.

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Shing Jeng, Doctor, Principal Investigator — Department of Neurology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Lindenberg R, Renga V, Zhu LL, Nair D, Schlaug G. Bihemispheric brain stimulation facilitates motor recovery in chronic stroke patients. Neurology. 2010 Dec 14;75(24):2176-84. doi: 10.1212/WNL.0b013e318202013a. Epub 2010 Nov 10. PMID 21068427
- [Background] Hesse S, Waldner A, Mehrholz J, Tomelleri C, Pohl M, Werner C. Combined transcranial direct current stimulation and robot-assisted arm training in subacute stroke patients: an exploratory, randomized multicenter trial. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):838-46. doi: 10.1177/1545968311413906. Epub 2011 Aug 8. PMID 21825004
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Stagg CJ, Bachtiar V, O'Shea J, Allman C, Bosnell RA, Kischka U, Matthews PM, Johansen-Berg H. Cortical activation changes underlying stimulation-induced behavioural gains in chronic stroke. Brain. 2012 Jan;135(Pt 1):276-84. doi: 10.1093/brain/awr313. Epub 2011 Dec 6. PMID 22155982
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Weiss T, Sens E, Teschner U, Meissner W, Preul C, Witte OW, Miltner WH. Deafferentation of the affected arm: a method to improve rehabilitation? Stroke. 2011 May;42(5):1363-70. doi: 10.1161/STROKEAHA.110.601138. Epub 2011 Mar 31. PMID 21454817
- [Background] Ward NS, Cohen LG. Mechanisms underlying recovery of motor function after stroke. Arch Neurol. 2004 Dec;61(12):1844-8. doi: 10.1001/archneur.61.12.1844. PMID 15596603
- [Derived] Koh CL, Lin JH, Jeng JS, Huang SL, Hsieh CL. Effects of Transcranial Direct Current Stimulation With Sensory Modulation on Stroke Motor Rehabilitation: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Dec;98(12):2477-2484. doi: 10.1016/j.apmr.2017.05.025. Epub 2017 Jun 24. PMID 28652065